CLINICAL TRIAL: NCT00756275
Title: Varenicline and Motivational Advice for Smokers With SUD
Brief Title: Varenicline and Motivational Advice for Smokers With Substance Use Disorders
Acronym: VARSUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Damaris J. Rohsenow, Ph.D., Professor (Research): Behavioral and Social Sciences, Brown University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01DA024652 (NIH); R01DA024652 (NIH)
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Results first posted 2018-05-08 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Smoking Cessation; Nicotine Dependence
Keywords: Tobacco Smoking; Smoking Cessation; Nicotine Dependence; Tobacco Use Disorder
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder; Tobacco Smoking | interventions — Nicotine Replacement Therapy; Varenicline; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicotine Replacement + PLA pill (Active Comparator): Nicotine replacement treatment patch plus matched placebo pill
  Interventions: Drug: Nicotine Replacement Treatment (NRT); Behavioral: Behavioral counseling for smoking cessation
- Varenicline + PLA patch (Active Comparator): Varenicline plus matched placebo patches containing no nicotine
  Interventions: Drug: varenicline; Behavioral: Behavioral counseling for smoking cessation

INTERVENTIONS:
Drug: Nicotine Replacement Treatment (NRT) — Nicotine replacement treatment (NRT) will follow the clinical practice guidelines for nicotine patch for people smoking at least 10 cigarettes per day (USDHHS, 2000), modified to allow 12 weeks use (tapering recommended for people with AUDs by Hughes et al., 2003b): 21 mg/day for 4 weeks, 14 mg/day for 4 weeks, 7 mg/day for 4 weeks.
  Other Names: Nicotine replacement therapy; Nicotine replacement treatment; NRT
  Arms: Nicotine Replacement + PLA pill
Drug: varenicline — Varenicline (VAR, 2 mg/d in divided doses) will be administered as follows. VAR: participant takes 0.5 mg/d for the first 3 days, 1 mg/d (0.5 mg 2x/d) for the next 4 days, and 2mg/d (1.0mg 2x/d) for 12 weeks.
  Other Names: VAR; Chantix
  Arms: Varenicline + PLA patch
Behavioral: Behavioral counseling for smoking cessation — The counseling consists of 10 sessions of Brief Advice (BA).BA is a simple smoking cessation counseling strategy: Assess smoking and initial interest in cessation, advise patient to quit smoking, assist patient in quitting, discussion of sobriety specific concerns, and cognitive-behavioral skills training. Medication management is conducted in every session, smoking cessation pamphlets are available. Session 1 (60 min, in-person) will be 1 week before Quit Day.Session 2 (30 min, in-person) takes place on Quit Day. Session 3 (10 min, in-person) will be 1 week later. Sessions 4-10 will be 5-10 min. telephone contacts at Weeks 2, 3, 4, 6, 8, 10, and 12 after Quit Day.
  Other Names: Behavioral treatment for smoking cessation; Behavioral counseling for quitting; Behavioral treatment for quitting

SUMMARY:
The purpose of this study is to evaluate the effects of 12 weeks of varenicline as compared to nicotine replacement therapy for smoking cessation among outpatients in treatment for substance use disorders. The intervention also incorporates counseling (Brief Advice), (adapted for sobriety settings), skills training and medication management.

DETAILED DESCRIPTION:
People with substance use disorders (SUD) have a high prevalence and rate of smoking with little success in quitting, so stronger approaches are needed to encourage attempts to quit smoking. Brief advice (BA), to motivate cessation, produced some benefit but low abstinence rates for smokers with SUDs while adding free transdermal nicotine replacement therapy (NRT) improved short-term cessation rates. Varenicline has been found to produce higher rates of short and long-term abstinence than bupropion or placebo. However, a comparison between the efficacy of varenicline and NRT has not yet conducted with people with SUDs. Given the lack of effectiveness for standard smoking treatments for this population, what needs to be known is whether varenicline would increase the smoking abstinence rates relative to NRT when all receive motivational counseling.

The primary aim of this study is to evaluate the effects of 12 weeks of varenicline as compared to NRT, using a two-group randomized placebo-controlled design on smoking cessation rates for 12 months among 274 outpatients in treatment for SUD. The counseling incorporates BA (adapted slightly for sobriety settings by directly addressing barriers and concerns expressed by substance abusers), skills training and medication management. Confirmed point-prevalence and sustained abstinence will be assessed at 3 and 6 a months after the start of treatment. Secondary aims will examine potential mediators of effect including within-treatment abstinence, craving, and nicotine withdrawal levels.

The potential significance is to add to knowledge about the most effective ways to maximize smoking cessation among substance abusers, important given that no methods are known to work with this difficult population. No study published to date has compared varenicline to NRT for efficacy with patients with SUD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of substance abuse or dependence by DSM-IV criteria
* Currently smoking at least 10 cigarettes per day for the past 6 months

Exclusion Criteria:

* Active psychosis or marked organic impairment according to medical records, or evidence of hallucinations or delusions
* Current use of any nicotine replacement, or other smoking cessation treatment
* Medical contraindications for NRT (including pregnancy, nursing, women not using birth control during heterosexual sex, history of unstable angina, history of severe congestive heart failure, uncontrolled hypertension, lung cancer, supplemental oxygen, allergy to adhesive, severe skin disease that requires treatment)
* Medical contraindications for VAR (including pregnancy, nursing, severe renal impairment by laboratory test, history of intolerance of varenicline, history of serious suicidal ideation or attempts in the past 5 years)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2009-01; Primary Completion 2014-03 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damaris J Rohsenow, Ph.D., Principal Investigator — Brown University; Rosemarie Martin, Ph.D., Study Director — Brown University
Locations (1):
- Brown University, Center for Alcohol and Addiction Studies, Providence, Rhode Island, United States

REFERENCES:
- [Background] Stapleton JA, Watson L, Spirling LI, Smith R, Milbrandt A, Ratcliffe M, Sutherland G. Varenicline in the routine treatment of tobacco dependence: a pre-post comparison with nicotine replacement therapy and an evaluation in those with mental illness. Addiction. 2008 Jan;103(1):146-54. doi: 10.1111/j.1360-0443.2007.02083.x. Epub 2007 Nov 19. PMID 18028247
- [Background] Rohsenow DJ, Monti PM, Colby SM, Martin RA. Brief interventions for smoking cessation in alcoholic smokers. Alcohol Clin Exp Res. 2002 Dec;26(12):1950-1. doi: 10.1097/01.ALC.0000041006.59547.9A. No abstract available. PMID 12500132
- [Result] Rohsenow DJ, Tidey JW, Martin RA, Colby SM, Swift RM, Leggio L, Monti PM. Varenicline versus nicotine patch with brief advice for smokers with substance use disorders with or without depression: effects on smoking, substance use and depressive symptoms. Addiction. 2017 Oct;112(10):1808-1820. doi: 10.1111/add.13861. Epub 2017 Jul 4. PMID 28498504
- [Result] Murphy CM, MacKillop J, Martin RA, Tidey JW, Colby SM, Rohsenow DJ. Effects of varenicline versus transdermal nicotine replacement therapy on cigarette demand on quit day in individuals with substance use disorders. Psychopharmacology (Berl). 2017 Aug;234(16):2443-2452. doi: 10.1007/s00213-017-4635-4. Epub 2017 May 13. PMID 28500373

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Five individuals enrolled were found to not meet study criteria, 3 did not pass the medical screen, and 13 individuals were lost prior to being randomized.
Groups:
- Nicotine Replacement + PLA Pill: Nicotine replacement treatment (NRT) patch plus matched placebo pill
  NRT will follow the clinical practice guidelines for people smoking at least 10 cigarettes per day (USDHHS, 2000), modified to allow 12 weeks use: 21mg/day for 4 weeks, 14mg/day for 4 weeks, 7mg/day for 4 weeks.
  Behavioral counseling for smoking cessation consists of 10 sessions of Brief Advice (BA).BA is a simple smoking cessation counseling strategy: Assess smoking and initial interest in cessation, advise patient to quit smoking, assist patient in quitting, discussion of sobriety specific concerns, and cognitive-behavioral skills training. Medication management is conducted in every session, smoking cessation pamphlets are available. Session 1 (60 min, in-person) will be 1 week before Quit Day.Session 2 (30 min, in-person) takes place on Quit Day. Session 3 (10 min, in-person) will be 1 week later. Sessions 4-10 will be 5-10 min. telephone contacts at Weeks 2, 3, 4, 6, 8, 10, and 12 after quit day.
- Varenicline + PLA Patch: Varenicline plus matched placebo patches containing no nicotine
  varenicline: Varenicline (VAR, 2mg/d in divided doses) will be administered as follows. VAR: participant takes 0.5 mg/d for the first 3 days, 1 mg/d (0.5 mg 2x/d) for the next 4 days, and 2mg/d (1.0mg 2x/d) for 12 weeks.
  Behavioral counseling for smoking cessation consists of 10 sessions of Brief Advice (BA).BA is a simple smoking cessation counseling strategy: Assess smoking and initial interest in cessation, advise patient to quit smoking, assist patient in quitting, discussion of sobriety specific concerns, and cognitive-behavioral skills training. Medication management is conducted in every session, smoking cessation pamphlets are available. Session 1 (60 min, in-person) will be 1 week before Quit Day.Session 2 (30 min, in-person) takes place on Quit Day. Session 3 (10 min, in-person) will be 1 week later. Sessions 4-10 will be 5-10 min. telephone contacts at Weeks 2, 3, 4, 6, 8, 10, and 12 after quit day.
Period: Overall Study
Arm/Group | Nicotine Replacement + PLA Pill | Varenicline + PLA Patch
Started | 60 | 77
Completed | 31 | 49
Not Completed | 29 | 28
Not completed — Lost to Follow-up | 25 | 21
Not completed — Withdrawal by Subject | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Nicotine Replacement + PLA Pill: Nicotine Replacement Treatment (NRT): Nicotine replacement treatment (NRT) will follow the clinical practice guidelines for nicotine patch for people smoking at least 10 cigarettes per day (USDHHS, 2000), modified to allow 12 weeks use (tapering recommended for people with AUDs by Hughes et al., 2003b): 21 mg/day for 4 weeks, 14 mg/day for 4 weeks, 7 mg/day for 4 weeks.
  Behavioral counseling for smoking cessation consists of 10 sessions of Brief Advice (BA).BA is a simple smoking cessation counseling strategy: Assess smoking and initial interest in cessation, advise patient to quit smoking, assist patient in quitting, discussion of sobriety specific concerns, and cognitive-behavioral skills training. Medication management is conducted in every session, smoking cessation pamphlets are available. Session 1 (60 min, in-person) will be 1 week before Quit Day.Session 2 (30 min, in-person) takes place on Quit Day. Session 3
- Varenicline + PLA Patch: varenicline: Varenicline (VAR, 2 mg/d in divided doses) will be administered as follows. VAR: participant takes 0.5 mg/d for the first 3 days, 1 mg/d (0.5 mg 2x/d) for the next 4 days, and 2mg/d (1.0mg 2x/d) for 12 weeks.
  Behavioral counseling for smoking cessation consists of 10 sessions of Brief Advice (BA).BA is a simple smoking cessation counseling strategy: Assess smoking and initial interest in cessation, advise patient to quit smoking, assist patient in quitting, discussion of sobriety specific concerns, and cognitive-behavioral skills training. Medication management is conducted in every session, smoking cessation pamphlets are available. Session 1 (60 min, in-person) will be 1 week before Quit Day.Session 2 (30 min, in-person) takes place on Quit Day. Session 3 (10 min, in-person) will be 1 week later. Sessions 4-10 will be 5-10 min. telephone contacts at Weeks 2, 3, 4, 6, 8, 10, and 12 after Quit Day.
  Pl
- Total: Total of all reporting groups
Arm/Group | Nicotine Replacement + PLA Pill | Varenicline + PLA Patch | Total
Number analyzed (Participants) | 60 | 77 | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 77 | 137
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.20 (9.7) | 39.96 (10.51) | 39.6 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 38 | 65
  Male | 33 | 39 | 72
Region of Enrollment [Number; unit: participants]
  United States | 60 | 77 | 137

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point-prevalence Smoking Abstinence
Description: 7 -day smoking cessation confirmed by expired alveolar CO levels of < 10 ppm or salivary cotinine < 16 ng/ml.
Time Frame: 3 month follow up
Population: "Intent to Treat" Note: People who were lost were counted as smoked
Measure: Number; unit: participants
Groups:
- Nicotine Replacement + PLA Pill: Nicotine replacement treatment (NRT) patch plus matched placebo pill
  NRT will follow the clinical practice guidelines for people smoking at least 10 cigarettes per day (USDHHS, 2000), modified to allow 12 weeks use : 21 mg/day for 4 weeks, 14 mg/day for 4 weeks, 7 mg/day for 4 weeks.
  Behavioral counseling for smoking cessation consists of 10 sessions of Brief Advice (BA).BA is a simple smoking cessation counseling strategy: Assess smoking and initial interest in cessation, advise patient to quit smoking, assist patient in quitting, discussion of sobriety specific concerns, and cognitive-behavioral skills training. Medication management is conducted in every session, smoking cessation pamphlets are available. Session 1 (60 min, in-person) will be 1 week before Quit Day.Session 2 (30 min, in-person) takes place on Quit Day. Session 3 (10 min, in-person) will be 1 week later. Sessions 4-10 will be 5-10 min. telephone contacts at Weeks 2, 3, 4, 6, 8, 10, and 12 after quit day.
- Varenicline + PLA Patch: Varenicline plus matched placebo patches containing no nicotine
  Varenicline (VAR, 2 mg/d in divided doses) will be administered as follows. VAR: participant takes 0.5 mg/d for the first 3 days, 1 mg/d (0.5 mg 2x/d) for the next 4 days, and 2mg/d (1.0mg 2x/d) for 12 weeks.
  Behavioral counseling for smoking cessation consists of 10 sessions of Brief Advice (BA).BA is a simple smoking cessation counseling strategy: Assess smoking and initial interest in cessation, advise patient to quit smoking, assist patient in quitting, discussion of sobriety specific concerns, and cognitive-behavioral skills training. Medication management is conducted in every session, smoking cessation pamphlets are available. Session 1 (60 min, in-person) will be 1 week before Quit Day.Session 2 (30 min, in-person) takes place on Quit Day. Session 3 (10 min, in-person) will be 1 week later. Sessions 4-10 will be 5-10 min. telephone contacts at Weeks 2, 3, 4, 6, 8, 10, and 12 after quit day.
Arm/Group | Nicotine Replacement + PLA Pill | Varenicline + PLA Patch
Number analyzed (Participants) | 60 | 77
participants | 2 | 10
Statistical Analysis 1: Comparison: Nicotine Replacement + PLA Pill vs Varenicline + PLA Patch; Test type: Superiority or Other; p < 0.05, Chi-squared; Odds Ratio (OR) = 4.33, 95% CI 2-sided [.91 to 20.56]

2. Secondary Outcome: Length of Longest Continuous Abstinence
Time Frame: Weeks 9 to 12
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Nicotine Replacement + PLA Pill | Varenicline + PLA Patch
Number analyzed (Participants) | 60 | 77
Days | 6.25 (10.06) | 7.84 (11.39)
Statistical Analysis 1: Comparison: Nicotine Replacement + PLA Pill vs Varenicline + PLA Patch; Test type: Superiority or Other; p = .50, t-test, 2 sided; Mean Difference (Final Values) = -1.59, 95% CI 2-sided [-6.29 to 3.11], Standard Error of Mean 2.36

3. Primary Outcome: 7-day Point-prevalence Smoking Abstinence
Description: 7 -day smoking cessation confirmed by expired alveolar CO levels of < 10 ppm or salivary cotinine < 16 ng/ml.
Time Frame: 6 month follow up
Measure: Number; unit: participants
Arm/Group | Nicotine Replacement + PLA Pill | Varenicline + PLA Patch
Number analyzed (Participants) | 60 | 77
participants | 2 | 7
Statistical Analysis 1: Comparison: Nicotine Replacement + PLA Pill; Test type: Superiority or Other; p = .30, Fisher Exact; Odds Ratio (OR) = 2.90, 95% CI 2-sided [.58 to 14.50]

4. Secondary Outcome: Percent Smoking Days
Time Frame: 3 month follow up
Population: Outcome data available for 89 participants who completed 3 month follow up.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Nicotine Replacement + PLA Pill | Varenicline + PLA Patch
Number analyzed (Participants) | 37 | 52
percentage of days | 62.39 (38.84) | 70.37 (38.79)
Statistical Analysis 1: Comparison: Nicotine Replacement + PLA Pill vs Varenicline + PLA Patch; Test type: Superiority or Other; p = .34, t-test, 2 sided; Mean Difference (Final Values) = -7.98, 95% CI 2-sided [-24.64 to 8.68], Standard Error of Mean 8.38

5. Secondary Outcome: Percent Smoking Days
Time Frame: 6 month follow up
Population: Outcome data available for 80 participants who completed 6 month follow up.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Nicotine Replacement + PLA Pill | Varenicline + PLA Patch
Number analyzed (Participants) | 31 | 49
percentage of days | 84.52 (31.25) | 77.12 (37.61)
Statistical Analysis 1: Comparison: Nicotine Replacement + PLA Pill vs Varenicline + PLA Patch; Test type: Superiority or Other; p = .36, t-test, 2 sided; Mean Difference (Final Values) = 7.39, 95% CI 2-sided [-8.73 to 23.52], Standard Error of Mean 8.10

6. Secondary Outcome: Percent Relapsed to Drug Use
Time Frame: 3 month follow up
Population: Outcome data available for 89 participants who completed 3 month follow up.
Measure: Number; unit: percentage of participants
Arm/Group | Nicotine Replacement + PLA Pill | Varenicline + PLA Patch
Number analyzed (Participants) | 37 | 52
percentage of participants | 12 | 14
Statistical Analysis 1: Comparison: Nicotine Replacement + PLA Pill vs Varenicline + PLA Patch; Test type: Superiority or Other; p = .57, Chi-squared

7. Secondary Outcome: Percent Relapsed to Drug Use
Time Frame: 6 month follow up
Population: Outcome data available for 80 participants who completed 6 month follow up.
Measure: Number; unit: percentage of participants
Arm/Group | Nicotine Replacement + PLA Pill | Varenicline + PLA Patch
Number analyzed (Participants) | 31 | 49
percentage of participants | 8 | 18
Statistical Analysis 1: Comparison: Nicotine Replacement + PLA Pill vs Varenicline + PLA Patch; Test type: Superiority or Other; p = .31, Chi-squared

8. Secondary Outcome: Percent Relapsed to Any Heavy Drinking
Description: 6 or more drinks for men; 5 or more drinks for women
Time Frame: 3 month follow up
Population: Outcome data available for 89 participants who completed 3 month follow up.
Measure: Number; unit: percentage of participants
Arm/Group | Nicotine Replacement + PLA Pill | Varenicline + PLA Patch
Number analyzed (Participants) | 37 | 51
percentage of participants | 7 | 9
Statistical Analysis 1: Comparison: Nicotine Replacement + PLA Pill vs Varenicline + PLA Patch; Test type: Superiority or Other; p = .72, Chi-squared

9. Secondary Outcome: Percent Relapsed to Any Heavy Drinking
Description: 6 or more drinks for men; 5 or more drinks for women
Time Frame: 6 month follow up
Population: Outcome data available for 80 participants who completed 6 month follow up.
Measure: Number; unit: percentage of particpiants
Arm/Group | Nicotine Replacement + PLA Pill | Varenicline + PLA Patch
Number analyzed (Participants) | 31 | 49
percentage of particpiants | 9 | 8
Statistical Analysis 1: Comparison: Nicotine Replacement + PLA Pill vs Varenicline + PLA Patch; Test type: Superiority or Other; p = .18, Chi-squared

10. Secondary Outcome: Beck Depression Inventory
Description: 0-10 = These ups and downs are considered normal 11-16 = Mild mood disturbance 17-20 = Borderline clinical depression 21-30 = Moderate depression 31-40 = Severe depression over 40 = Extreme depression
Time Frame: Week 12
Population: Outcome data available for 80 participants who had valid depression data 12 week assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nicotine Replacement + PLA Pill | Varenicline + PLA Patch
Number analyzed (Participants) | 36 | 44
units on a scale | 5.19 (6.53) | 5.75 (8.47)
Statistical Analysis 1: Comparison: Nicotine Replacement + PLA Pill vs Varenicline + PLA Patch; Test type: Superiority or Other; p = .75, t-test, 2 sided; Mean Difference (Final Values) = -.56, 95% CI 2-sided [-3.98 to 2.87], Standard Error of Mean 1.72

ADVERSE EVENTS:
Description: Structured interviews weekly for 12 weeks and at 3 & 6 months and as reported any time by participant or clinical staff member.
Arm/Group | Nicotine Replacement + PLA Pill | Varenicline + PLA Patch
Serious Adverse Events (participants affected / at risk) | 3/60 | 10/77
Other Adverse Events (participants affected / at risk) | 3/60 | 1/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Replacement + PLA Pill (N=60) | Varenicline + PLA Patch (N=77)
substance abuse (hospital or death) (Psychiatric disorders) | 1 (1) | 4 (4)
accidents (ER or hospital) (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
hospital and respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (7) | 0 (0)
pregnancy complication (Reproductive system and breast disorders) | 0 (0) | 1 (1)
diabetic complication (Endocrine disorders) | 0 (0) | 1 (1)
disorientation (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Replacement + PLA Pill (N=60) | Varenicline + PLA Patch (N=77)
increased depression (Psychiatric disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No